CLINICAL TRIAL: NCT06894979
Title: A Phase I Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of AZD1390 (NSC# 852149) When Combined With Focal Radiation in Pediatric Patients With High Grade Glioma
Brief Title: Testing the Addition of an Anti-Cancer Drug, AZD1390, During Radiation Therapy for Newly Diagnosed High Grade Glioma, Diffuse Midline Glioma, or Diffuse Intrinsic Pontine Glioma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEPN2415; NCI-2025-01429 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PEPN2415 (Other: Pediatric Early Phase Clinical Trial Network); PEPN2415 (Other: CTEP); UM1CA228823 (NIH)
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-06

CONDITIONS: Childhood Astrocytoma; Childhood Diffuse Intrinsic Pontine Glioma; Childhood Diffuse Midline Glioma; Childhood Glioblastoma; Childhood Malignant Glioma
MeSH Terms: conditions — Astrocytoma | interventions — AZD1390; Specimen Handling; Magnetic Resonance Spectroscopy; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (AZD1390 and radiation therapy) (Experimental): Patients receive AZD1390 PO once within 5 days prior to radiation therapy. Patients then receive AZD1390 PO QD, 5 days per week, Monday through Friday, and also receive radiation therapy on the same days for approximately 6 weeks. Patients then receive AZD1390 on days 1-14 after radiation in the absence of disease progression or unacceptable toxicity. Patients undergo MRI and blood sample collection and may optionally undergo cerebrospinal fluid collection throughout the study.
  Interventions: Drug: ATM Kinase Inhibitor AZD1390; Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Radiation: Radiation Therapy; Other: Survey Administration

INTERVENTIONS:
Drug: ATM Kinase Inhibitor AZD1390 — Given PO
  Other Names: AZD-1390; AZD1390
Procedure: Biospecimen Collection — Undergo blood and cerebrospinal fluid collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Other: Survey Administration — Ancillary studies

SUMMARY:
This phase I clinical trial studies the side effects and best dose of AZD1390 and to see how well it works when given together with radiation therapy for the treatment of pediatric patients with high grade glioma, diffuse midline glioma or diffuse intrinsic pontine glioma. AZD1390 is in a class of medications called kinase inhibitors. It works by blocking the signals that cause cancer cells to multiply. This helps to stop the spread of cancer cells. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill cancer cells and shrink tumors. Giving AZD1390 with radiation may be safe, tolerable, and/or effective in treating pediatric patients with high grade glioma, diffuse midline glioma or diffuse intrinsic pontine glioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define the recommended phase 2 dose of ATM Kinase Inhibitor AZD1390 (AZD1390) when given in combination with radiation for pediatric supratentorial high-grade gliomas.

II. To define the recommended phase 2 dose of AZD1390 when given in combination with radiation for pediatric infratentorial high-grade gliomas.

III. To define the toxicities and characterize the safety profile of AZD1390 when given in combination with radiation for pediatric supratentorial high-grade gliomas.

IV. To define the toxicities and characterize the safety profile of AZD1390 when given in combination with radiation for pediatric infratentorial high-grade gliomas.

V. To characterize the pharmacokinetic profile of AZD1390 when given in combination with radiation to pediatric patients for pediatric supratentorial and infratentorial high-grade gliomas.

SECONDARY OBJECTIVES:

I. To evaluate preliminary efficacy when AZD1390 is given in combination with radiation to pediatric patients with supratentorial high-grade gliomas as determined via progression free survival (PFS), overall survival (OS) and overall radiographic response (ORR) within the confines of a phase 1 trial.

II. To evaluate preliminary efficacy when AZD1390 is given in combination with radiation to pediatric patients with infratentorial high-grade gliomas as determined via PFS, OS and ORR within the confines of a phase 1 trial.

III. To obtain preliminary data on neurological function of patients with supratentorial and infratentorial high-grade gliomas receiving AZD1390 and focal radiation via the pediatric neurologic assessment in neuro-oncology (NANO) scale.

EXPLORATORY OBJECTIVES:

I. To evaluate changes in neurocognitive function from baseline (within 2 weeks of enrollment) to end of protocol directed therapy (completion of AZD1390), at 22 weeks (5.5 months) and at 44 weeks (11.5 months) after completion of radiation.

II. To evaluate changes in patient reported outcomes utilizing Patient Reported Outcomes Measurement Information System (PROMIS) from baseline (within 2 weeks of enrollment) and at the time of imaging assessments.

III. To evaluate the alternative lengthening of telomeres (ALT) phenotype in archival tumor and cell-free deoxyribonucleic acid (cfDNA) in patients with high grade glioma (HGG) undergoing AZD1390 and radiation therapy.

IV. To evaluate the correlation of genomic, transcriptomic, proteomic, and cytokine markers, including homologous recombination deficiency (HRD) and associated mutational signatures and TP53/related DNA repair gene mutational status, with response to AZD1390 and radiation therapy.

V. Evaluate differences in radiation dosimetry to organs at risk and target volumes by radiation technique and modality and its correlation with toxicity and response and survival.

VI. Evaluate cfDNA in plasma and cerebrospinal fluid (CSF) (when obtained) and pharmacodynamic markers of peripheral blood mononuclear cells (PBMCs) prior, during and after therapy to better understand its correlation with treatment response.

OUTLINE: This is a dose-escalation study of AZD1390 in combination with radiation.

Patients receive AZD1390 orally (PO) once within 5 days prior to radiation therapy. Patients then receive AZD1390 PO once daily (QD), 5 days per week, Monday through Friday, and also receive radiation therapy on the same days for approximately 6 weeks. Patients then receive AZD1390 on days 1-14 after radiation in the absence of disease progression or unacceptable toxicity. Patients undergo magnetic resonance imaging (MRI) and blood sample collection and may optionally undergo cerebrospinal fluid collection throughout the study.

After completion of study treatment, patients are followed up at 30 days and then every 8 weeks until progression or 2 years after the last dose of AZD1390 as well as at 22 and 44 weeks after completion of radiation therapy. From progression, patients are followed up will be every 6 months until year 4 from the last dose of AZD1390 then yearly until year 5.

ELIGIBILITY:
Inclusion Criteria:

* COHORT A and COHORT B: For the dose escalation phase, patients must be ≥ 12 months and < 18 years of age at the time of study enrollment
* COHORT C and COHORT D: For the disease expansion phase, patients must be ≥ 12 months and < 22 years of age at the time of study enrollment
* Patients with newly diagnosed primary high-grade glioma (HGG), diffuse midline glioma (DMG) (excluding primary spinal tumors), or diffuse intrinsic pontine glioma (DIPG) who are eligible to receive 54-59.4 grey (Gy) fractionated radiation at 1.8 Gy/day. Patients must have had histologic verification of malignancy at original diagnosis except in patients with DIPG as defined below.

  * COHORTS A AND C (SUPRATENTORIAL TUMORS):

    * HGG and non-pontine DMG:

      * Patients with newly diagnosed HGG (including diffuse hemispheric glioma, H3 G34-mutant; diffuse pediatric-type high-grade glioma, H3-wildtype and IDH-wildtype; astrocytoma; IDH-mutant; or glioblastoma, IDH-wildtype): or non-pontine DMG (including diffuse midline glioma, H3 K27-altered; diffuse pediatric-type high-grade glioma, H3-wildtype and IDH-wildtype; astrocytoma; IDH-mutant; or glioblastoma, IDH-wildtype) require histologic diagnosis.
  * COHORT B AND D (INFRATENTORIAL TUMORS):

    * DIPG/pontine DMG or infratentorial HGG or DMG:

      * Patients with newly diagnosed typical DIPG, defined as tumors with a pontine epicenter and diffuse involvement of at least 2/3 of the pons on at least 1 axial T2-weighted image, are eligible. No histologic confirmation is required.
      * Patients with infratentorial tumors that do not meet radiographic criteria for typical DIPG (e.g., focal tumors or those involving less than 2/3 of the pontine cross-sectional area with or without extrapontine extension) are eligible if the tumors are biopsied and proven to be high-grade gliomas (including diffuse midline glioma H3 K27-altered; diffuse pediatric-type high-grade glioma, H3-wildtype and IDH-wildtype; astrocytoma; IDH-mutant; or glioblastoma, IDH-wildtype) by institutional diagnosis.
  * Protocol Definitions

    * Supratentorial tumors are defined as tumors with an epicenter in the cerebral hemispheres, basal ganglia, thalamus, hypothalamus, or pituitary gland.
    * Infratentorial tumors are defined as tumors with an epicenter in the brainstem, cerebellum
* Patients with measurable or non-measurable (following a gross total resection) disease
* Karnofsky ≥ 50% for patients > 16 year of age and Lansky ≥ 50% for patients ≤ 16 years of age.

  * Note: Patients who are unable to walk because of paralysis, but who are in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Prior therapy for any cancer diagnosis (including radiation) is not allowed with the exception of surgery and/or corticosteroids. If receiving corticosteroids, dose must remain stable or decrease after enrollment
* Peripheral absolute neutrophil count (ANC) ≥ 1000/uL (must be performed within 7 days prior to enrollment unless otherwise indicated)
* Platelet count ≥ 100,000/uL (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment) (must be performed within 7 days prior to enrollment unless otherwise indicated)
* Hemoglobin ≥ 8.0 g/dL at baseline (may receive red blood cell [RBC] transfusions) (must be performed within 7 days prior to enrollment unless otherwise indicated)
* A creatinine based on age/sex as follows (must be performed within 7 days prior to enrollment unless otherwise indicated):

  * 1 to < 2 years: Maximum serum creatinine 0.6 mg/dL (male), 0.6 mg/dL (female)
  * 2 to < 6 years: Maximum serum creatinine 0.8 mg/dL (male), 0.8 mg/dL (female)
  * 6 to < 10 years: Maximum serum creatinine 1 mg/dL (male), 1 mg/dL (female)
  * 10 to < 13 years: Maximum serum creatinine 1.2 mg/dL (male), 1.2 mg/dL (female)
  * 13 to < 16 years: Maximum serum creatinine 1.5 mg/dL (male), 1.4 mg/dL (female)
  * >= 16 years: Maximum serum creatinine 1.7 mg/dL (male),1.4 mg/dL (female) OR a 24 hour urine creatinine clearance ≥ 70 mL/min/1.73 m^2 OR a glomerular filtration rate (GFR) ≥ 70 mL/min/1.73 m^2. GFR must be performed using direct measurement with a nuclear blood sampling method OR direct small molecule clearance method (iothalamate or other molecule per institutional standard).

Note: Estimated GFR (eGFR) from serum creatinine, cystatin C or other estimates are not acceptable for determining eligibility

* Note: The threshold creatinine values in this Table were derived from the Schwartz formula for estimating GFR (Schwartz et al. J. Peds, 106:522, 1985) utilizing child length and stature data published by the CDC.

  * Bilirubin (sum of conjugated + unconjugated or total) ≤ 1.5 x upper limit of normal (ULN) for age except in patients diagnosed with Gilbert's disease for which bilirubin must be ≤ 3.0 × ULN (must be performed within 7 days prior to enrollment unless otherwise indicated)
  * Alanine aminotransferase (ALT) ≤ 3 x ULN, unless attributed to tumor involvement then ALT ≤ 5 x ULN (must be performed within 7 days prior to enrollment unless otherwise indicated)
  * Aspartate aminotransferase (AST) ≤ 3 x ULN, unless attributed to tumor involvement then AST ≤ 5 x ULN (must be performed within 7 days prior to enrollment unless otherwise indicated)
  * Albumin ≥ 2 g/dL (must be performed within 7 days prior to enrollment unless otherwise indicated)
  * No evidence of dyspnea at rest, no exercise intolerance and a pulse oximetry > 93%
  * Patients with seizure disorder may be enrolled if on anticonvulsants and well controlled as evidenced by no increase in seizure frequency in the prior 7 days. If needed, evaluate use of enzyme-inducing anticonvulsants
  * Serum lipase ≤ 1.5 ULN (must be performed within 7 days prior to enrollment unless otherwise indicated)
  * Prothrombin time (PT)/international normalization rate (INR) < 1.5 x ULN (must be performed within 7 days prior to enrollment unless otherwise indicated)
  * Patients must have the ability to swallow whole tablets (AZD1390 may not be administered via nasogastric [NG]/gastric [G]-tubes)

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies, OR because there is yet no available information regarding human fetal or teratogenic toxicities. Pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use two effective methods of birth control, including a medically accepted barrier or contraceptive method (eg, male or female condom) for the duration of the study. Abstinence is an acceptable method of birth control. Women of childbearing potential should use adequate contraception during study participation and for 6 months after the last dose of AZD1390. Male patients with female partners of childbearing potential should use adequate contraception during study participation and for 16 weeks after the last dose of AZD1390
* Investigational Drugs: Patients who are currently receiving another investigational drug are not eligible
* Anti-cancer Agents: Patients who are currently receiving other anti-cancer agents are not eligible with the exception of corticosteroids
* Anti-graft versus host disease (GVHD) agents post-transplant: Patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial
* CYP-450/Transport Proteins: Patients receiving any medications or substances that are strong inhibitors or inducers of CYP3A4/5 enzyme are ineligible. Moderate inhibitors and inducers of CYP3A4/5 are permitted but caution should be exercised, and patients monitored closely for possible drug interactions. Strong inhibitors or inducers CYP3A4 should be stopped at least 2 weeks before the first dose of AZD1390 (3 weeks for St John's Wort). As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Enzyme-Inducing Anticonvulsants: Patients must not have received enzyme-inducing anticonvulsants within 14 days prior to enrollment
* Patients who have an uncontrolled infection are not eligible
* Patients who have received a prior solid organ transplantation are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible. This includes patients with rapidly declining neurological status
* Patients must have the ability to swallow whole tablets (AZD1390 may not be administered via NG/G-tubes). Patients with medical conditions that affect drug absorption, such as short gut syndrome are not eligible
* Patients with known macular degeneration, uncontrolled glaucoma, or cataracts are not eligible
* Patients with primary spinal cord high grade gliomas are not eligible
* Patients with metastatic disease are not eligible; Metastatic disease is defined as distant intracranial or spinal metastasis including leptomeningeal disease, or tumor cells within the CSF. MRI of the spine with and without contrast must be performed if metastatic disease is suspected by the treating physician
* Patients with gliomatosis type growth pattern (or diffuse spread) with involvement of at least 3 lobes of the brain are not eligible with the exception of H3 K27M-mutant bithalamic tumors
* Patients with infant-type hemispheric high-grade gliomas are excluded
* Patients with BRAFV600E mutations are excluded
* Patients who are not able to receive protocol specified radiation therapy
* Patients with a history of radiotherapy as part of anti-cancer therapy are excluded
* Presence of myopathy or raised CK > 5 x ULN on 2 occasions at screening will result in exclusion.

  * CK should not be measured following strenuous exercise or in the presence of a plausible alternative cause of CK increase, which may confound interpretation of the results.
  * If CK levels are significantly elevated at baseline (>5 x ULN) a confirmatory test should be carried out within 5 - 7 days.
  * If the repeat test confirms a baseline CK >5 x ULN, treatment should not be started
* HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible as long as they are NOT receiving anti-retroviral agents that are strong inhibitors or inducers of CYP3A4 or substrates of UGT1A1 and UGT1A9
* Evidence of clinically significant cardiac dysfunction or prolonged corrected QT interval (QTc) (> 450 msec) on baseline electrocardiogram (EKG)
* Patients with known hepatitis B or C with detectable viral load
* Any significant medical condition that in the medical judgement of the investigator would compromise the patient's ability to tolerate study drug or participate in the study

Ages: 12 Months to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) of ATM Kinase Inhibitor AZD1390 (AZD1390) for pediatric supratentorial high-grade gliomas | Up to 75 days
  The maximum tolerated dose or recommended phase 2 dose will be estimated by the isotonic estimates of toxicity probabilities for which the estimate of the DLT/RP2D rate is closed to the target rate of 25% in children and adolescents with supratentorial tumors.
Maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) of AZD1390 for pediatric infratentorial high-grade gliomas | Up to 75 days
  The maximum tolerated dose or recommended phase 2 dose will be estimated by the isotonic estimates of toxicity probabilities for which the estimate of the DLT/RP2D rate is closed to the target rate of 25% in children and adolescents with infratentorial tumors.
Incidence of adverse events for AZD1390 for pediatric supratentorial high-grade gliomas | Up to 5 years
  Frequency (%) of evaluable patients with toxicity at least possibly attributable to study agent stratified by study part and dose level using Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v 5.0).
Incidence of adverse events for AZD1390 for pediatric infratentorial high-grade gliomas | Up to 5 years
  Frequency (%) of evaluable patients with toxicity at least possibly attributable to study agent stratified by study part and dose level using Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v 5.0).
Maximum serum concentration of AZD1390 | Up to 24 hours
  Median (min, max) of the maximum serum concentration of AZD1390 assessed at time 0, 2, 4, 6, 8, and 24-hours post dose on cycle 1 day 1.
Time to peak drug concentration of AZD1390 | Up to 24 hours
  Median (min, max) of the time to peak drug concentration of AZD1390 assessed at time 0, 2, 4, 6, 8, and 24-hours post dose on cycle 1 day 1.
Elimination half-life of AZD1390 | Up to 24 hours
  Median (min, max) of the elimination half-life of AZD1390 assessed at time 0, 2, 4, 6, 8, and 24-hours post dose on cycle 1 day 1.
Clearance of AZD1390 | Up to 24 hours
  Median (min, max) of the clearance of AZD1390 assessed at time 0, 2, 4, 6, 8, and 24-hours post dose on cycle 1 day 1.
Volume of distribution of AZD1390 | Up to 24 hours
  Median (min, max) of the volume of distribution of AZD1390 assessed at time 0, 2, 4, 6, 8, and 24-hours post dose on cycle 1 day 1.

SECONDARY OUTCOMES:
Progression free survival (PFS) for patients with supratentorial high-grade gliomas | Up to 5 years
  Median (95% confidence interval) of the time to progression for patients with supratentorial high-grade gliomas.
Overall survival (OS) for patients with supratentorial high-grade gliomas | Up to 5 years
  Median (95% confidence interval) of the time to death due to any cause for patients supratentorial high-grade gliomas.
Overall radiographic response (ORR) for patients with supratentorial high-grade gliomas | Up to 5 years
  Best overall response (CR, PR, SD, PD) will be summarized by frequency (%) of response-evaluable patients with supratentorial high-grade gliomas.
PFS for patients with infratentorial high-grade gliomas | Up to 5 years
  Median (95% confidence interval) of the time to progression for patients with infratentorial high-grade gliomas.
OS for patients with infratentorial high-grade gliomas | Up to 5 years
  Median (95% confidence interval) of the time to death due to any cause for patients with supratentorial high-grade gliomas.
ORR for patients with infratentorial high-grade gliomas | Up to 5 years
  Best overall response (CR, PR, SD, PD) will be summarized by frequency (%) of response-evaluable patients with infratentorial high-grade gliomas.
Pediatric neurological assessment in neuro-oncology (pNANO) | Up to 5 years
  Median (min, max) pNANO scores stratified by disease cohort (supratentorial and infratentorial) and dose level at baseline and then every 8-weeks.

OTHER OUTCOMES:
Change in Neurocognitive function | Up to 44-weeks
  Median (min, max) change in scores for each of detection, identification, on-back, one-card learning, and Groton maze learning test stratified by disease cohort (supratentorial and infratentorial) and dose level at 22-weeks and 44-weeks versus baseline.
Change in patient reported outcomes measurement information system | Up to 5 years
  Median (min, max) change in PROMIS scores for each subdomain (Cognitive function, global health, 29 profile, early childhood parent report global health, and parent proxy every 8-weeks during the first 12-months and then every 3-4 months versus baseline.
Alternative lengthening of telomeres phenotype | Up to 5 days
  Frequency (%) of patients with alternative lengthening of telomeres (ALT) phenotype.
Genomic, transcriptomic, proteomic, and cytokine markers, including homologous recombination deficiency and associated mutational signatures and TP53/related deoxyribonucleic acid (DNA) repair gene mutational status | Up to 5 years
  Median (min, max) genomic, transcriptomic, proteomic, and cytoking markers stratified by patient best overall response.
Differences in radiation dosimetry to organs at risk and target volumes by radiation technique and modality | Up to 5 years
  Median (min, max) radiation dosimetry to organs at risk and target volumes by radiation technique and modality.
Circulating tumor DNA in plasma and CSF (when obtained) and pharmacodynamic markers of peripheral blood mononuclear cells | Up to 5 years
  Median (min, max) plasma ctDNA, CSF, and pharmacodynamic markers of PBMCs stratified by patient best overall response.

CONTACTS AND LOCATIONS:
Overall Officials: Erin K Barr, Principal Investigator — Pediatric Early Phase Clinical Trial Network
Locations (17):
- United States (17):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Seattle Children's Hospital, Seattle, Washington